CLINICAL TRIAL: NCT02418819
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED, PARALLEL GROUP, SPONSOR OPEN, PHASE 1B STUDY TO EXAMINE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF PF-06412562 IN PSYCHIATRICALLY STABLE SUBJECTS WITH SCHIZOPHRENIA
Brief Title: A Study To Examine Safety, Pharmacokinetics, And Pharmacodynamic Of Pf 06412562 In Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7441007
Record Dates: First submitted 2015-03-23; First posted 2015-04-16 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-06412562 3mg (Experimental): PF-06412562 3mg BID
  Interventions: Drug: PF-06412562 3mg BID
- PF-06412562 9mg (Experimental): PF-06412562 9mg BID
  Interventions: Drug: PF-06412562 9mg BID
- PF-06412562 45mg (Experimental): PF-06412562 45mg BID
  Interventions: Drug: PF-06412562 45mg BID
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06412562 3mg BID — PF-06412562
  Other Names: PF-06412562 3mg
  Arms: PF-06412562 3mg
Drug: PF-06412562 9mg BID — PF-06412562
  Other Names: PF-06412562 9mg
  Arms: PF-06412562 9mg
Drug: PF-06412562 45mg BID — PF-06412562
  Other Names: PF-06412562 45mg
  Arms: PF-06412562 45mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to investigate the safety, tolerability pharmacokinetics and pharmacodynamic effects of PF-06412562 following multiple dose administration as MR tablets in subjects with schizophrenia.

DETAILED DESCRIPTION:
B7441007 is a randomized, double-blind, placebo-controlled, sponsor open, parallel group design, Phase 1b study of the safety, tolerability, pharmacokinetics, and pharmacodynamics of 3 doses of PF-06412562 (3 mg BID, 9 mg BID and 45 mg BID) over 15 days in approximately 100 psychiatrically stable (as defined by the inclusion and exclusion criteria) subjects with schizophrenia are on background treatment with SOC antipsychotics and other psychotropic medications.

All doses will be administered twice daily, with approximately 12 hours between each dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with schizophrenia both male and female
2. Evidence of stable schizophrenia symptomatology for at least 3 months (no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of symptoms of schizophrenia, etc).
3. Subjects must be in ongoing maintenance antipsychotic therapy other than clozapine (oral or depot) on a stable medication treatment regimen for for at least 2 months prior to Day 1, including concomitant psychotropic medications.

Exclusion Criteria:

1. History of seizure
2. Pregnant or nursing females
3. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of screening and at the time of dosing).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Arcadia MRI & Imaging Center, Arcadia, California
  - California Clinical Trials Medical Group, Glendale, California
  - Glendale Adventist Medical Center, Glendale, California
  - Maryland Psychiatric Research Center (MPRC) of the University of Maryland, Baltimore, Maryland
  - CBH Health, LLC, Gaithersburg, Maryland
  - Foers Long Term Care Pharmacy LLC, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Arce E, Balice-Gordon R, Duvvuri S, Naylor M, Xie Z, Harel B, Kozak R, Gray DL, DeMartinis N. A novel approach to evaluate the pharmacodynamics of a selective dopamine D1/D5 receptor partial agonist (PF-06412562) in patients with stable schizophrenia. J Psychopharmacol. 2019 Oct;33(10):1237-1247. doi: 10.1177/0269881119855302. Epub 2019 Jul 2. PMID 31264510
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441007&StudyName=A%20Randomized%2C%20Double-blind%2C%20Placebo%20Controlled%2C%20Parallel%20Group%2C%20Sponsor%20Open%2C%20Phase%201b%20Study%20To%20Examine%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20Pf%2006412562%20In%20Psychiatrically%20Stable%20Subjects%20With%20Schizophrenia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 103 participants were randomized and assigned to study treatment. One (1) participant in the PF-06412562 3 mg twice a day (BID) group and 2 participants in the PF-06412562 45 mg BID group did not receive study drug. Therefore, 100 participants received study treatment.
Groups:
- PF-06412562 3 mg BID: Participant received 3 mg PF 06412562 modified release tablets were orally administered twice daily for 15 days with approximately 12 hours between each dose.
- PF-06412562 9 mg BID: Participant received 9 mg PF 06412562 modified release tablets were orally administered twice daily for 15 days with approximately 12 hours between each dose.
- PF-06412562 45 mg BID: Participant received 45 mg PF 06412562 modified release tablets were orally administered twice daily using a titration scheme (15 mg BID for 2 days, 30 mg BID for 2 days and 45 mg BID for the rest of the study) for 15 days with approximately 12 hours between each dose.
- Placebo: Participant received placebo matched to PF 06412562 3 mg and 15 mg modified release tablets were orally administered twice daily for 15 days with approximately 12 hours between each dose.
Period: Overall Study
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Started | 22 | 16 | 33 | 29
Completed | 21 | 16 | 29 | 28
Not Completed | 1 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 1 | 0
Not completed — No longer willing to participate | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo | Total
Number analyzed (Participants) | 22 | 16 | 33 | 29 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (6.1) | 34.3 (7.2) | 33.8 (6.9) | 35.7 (5.8) | 34.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 8 | 9 | 23
  Male | 19 | 13 | 25 | 20 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any events occurring following start of treatment or increasing in severity were counted as treatment emergent. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 7-10 days after last dose of study drug, up to 26 days
Population: The safety analysis set was used, defined as all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 33 | 29
Participants
  AEs | 10 | 10 | 17 | 14
  SAEs | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Supine and Standing Vital Signs Meeting Categorical Summarization Criteria
Description: Vital Signs tests included systolic and diastolic blood pressure (BP) and pulse rate of seated supine and standing . Vital signs categorical summarization criteria were 1), supine and standing BP: systolic (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from baseline, diastolic <50 mm Hg; 2), supine and standing pulse rate <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: Baseline up to 7-10 days after last dose of study drug, up to 26 days
Population: The safety analysis set was used, which defined as all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 33 | 29
Participants
  Supine SBP <90 mm Hg | 1 | 3 | 6 | 6
  Standing SBP <90 mm Hg | 1 | 0 | 1 | 1
  Supine DBP <50 mm Hg | 0 | 2 | 2 | 2
  Standing DBP <50 mm Hg | 0 | 0 | 0 | 0
  Supine Pulse rate <40 bpm | 0 | 0 | 0 | 0
  Supine Pulse rate >120 bpm | 0 | 0 | 0 | 0
  Standing Pulse rate <40 bpm | 0 | 0 | 0 | 0
  Standing Pulse rate >140 bpm | 0 | 0 | 0 | 0
  Increase: supine SBP >=30 mm Hg | 3 | 4 | 4 | 1
  Increase: standing SBP >=30 mm Hg | 1 | 1 | 0 | 3
  Increase: supine DBP >=20 mm Hg | 1 | 4 | 1 | 1
  Increase: standing DBP >=20 mm Hg | 0 | 0 | 0 | 2
  Decrease: supine SBP >= 30 mm Hg | 1 | 3 | 4 | 3
  Decrease: standing SBP >= 30 mm Hg | 2 | 0 | 2 | 2
  Decrease: supine DBP >=20 mm Hg | 3 | 3 | 9 | 5
  Decrease: standing DBP >=20 mm Hg | 2 | 1 | 1 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) (Standard 12-Lead) Data Meeting Categorical Summarization Criteria
Description: ECG categorical summarization criteria were 1), time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval): more than or equal to (>=) 200 milliseconds (msec); for percent change(PChg), >=25 percent (%) increase when baseline (b)>100 msec; or increase >=50% when b less than or equal to (<=)100 msec; 2), the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval): >=300 msec; >=25percent (%) increase when b >200 msec; or increase >=50% when b <=200 msec; 3), time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec and >=500 msec; increase from b >=30 - <60 and >=60 msec
Time Frame: Baseline up to 7-10 days after last dose of study drug, up to 26 days
Population: The safety analysis set was used, defined as all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 33 | 29
Participants
  PR interval >=300 msec | 0 | 0 | 0 | 0
  QRS complex >=200 msec | 0 | 0 | 0 | 0
  QTcF interval 450-480 msec | 0 | 0 | 1 | 0
  QTcF interval 480-500 msec | 0 | 0 | 0 | 0
  QTcF interval >=500 msec | 0 | 0 | 0 | 0
  PR interval increase b>200 & PChg>=25% | 0 | 0 | 0 | 0
  PR interval increase b<=200 & PChg>=50% | 0 | 0 | 0 | 0
  QRS complex increase b>100 & PChg>=25% | 0 | 0 | 0 | 0
  QRS complex increase b<=100 & PChg>=50% | 0 | 0 | 0 | 0
  QTcF interval increase 30-60 msec | 3 | 0 | 0 | 0
  QTcF interval increase >=60 msec | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Blood and Urine Safety Laboratory Test Abnormalities
Description: The total number of participants with blood and urine laboratory test abnormalities (without regard to baseline abnormality) was assessed. Clinical laboratory tests included hematology, chemistry, urinalysis, and some other tests.
Time Frame: Baseline up to Day 15
Population: The safety analysis set was used, defined as all participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 29 | 28
Participants | 9 | 8 | 8 | 12

5. Primary Outcome: Number of Participants With New Onset and Worsening of Post Baseline Suicidality in Columbia Suicide Severity Rating Scale (C-SSRS) on Day 1, Day 7 and Follow-up.
Description: The C-SSRS was an interview based rating scale to systematically assess suicidal ideation and suicidal behavior. Versions were available for Screening/Baseline and follow-up visits. Post-baseline suicidality was displayed without regard to baseline and as new onset or worsening relative to baseline. A participant was considered to have a new onset of suicidality if the participant reported no ideation and no behavior at the baseline assessment. A participant was considered to have a worsening of suicidality if the participant moved to a lower numbered Columbia Classification Algorithm of Suicide Assessment (C-CASA) category (observed in categories 1-4) than was reported at baseline.
Time Frame: Baseline, Days 1,7 and follow-up (7-10 days after last dose of study drug, up to 26 days)
Population: The safety analysis set was used, defined as all participants who received at least 1 dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 33 | 29
Participants
  Day1 New Onset | 0 | 0 | 0 | 0
  Day1 Worsening | 0 | 0 | 0 | 0
  Day7 New Onset | 0 | 0 | 0 | 0
  Day7 Worsening | 0 | 0 | 0 | 0
  Follow Up New Onset | 1 | 0 | 0 | 0
  Follow Up Worsening | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline to Day 13 of Wechsler Memory Scale (WMS III) Spatial Span + Letter Number Span Composite Score (Working Memory Domain)
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess working memory of participants. Total score range of this subset ranges from 40 (minimum score) to 60 (maximum score), with higher scores indicating better cognitive function.
Time Frame: Baseline, Day 13
Population: Per Protocol Analysis Set (PPAS)subset of Full Analysis Set(FAS).Criteria:1)Received all doses of study treatment to which they randomized2)No major protocol deviation3)Had baseline measurement and at least 1 post baseline measurement for at least 1 PD endpoint.Overall Number of Participants Analyzed=participants evaluable in this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 22 | 16 | 29 | 28
Scores on a scale | 3.95 (8.20) | 3.13 (7.90) | 1.28 (7.51) | 5.25 (6.96)
Statistical Analysis 1: Comparison: PF-06412562 3 mg BID vs Placebo; Baseline is defined as the Day -2 assessment; Test type: Superiority or Other; p = 0.8243, ANCOVA; One(1)-sided P-values were obtained from an ANCOVA model on change from baseline with baseline, treatment, site, gender and age as fixed effects; LSMean difference from placebo = -1.90, 92% CI 1-sided [lower limit -4.78], Standard Error of Mean 2.032
Statistical Analysis 2: Comparison: PF-06412562 9 mg BID vs Placebo; Baseline is defined as the Day -2 assessment; Test type: Superiority or Other; p = 0.8277, ANCOVA; One(1)-side P-values were obtained from an ANCOVA model on change from baseline with baseline, treatment, site, gender and age as fixed effects; LSMean difference from placebo = -2.14, 92% CI 1-sided [lower limit -5.33], Standard Error of Mean 2.252
Statistical Analysis 3: Comparison: PF-06412562 45 mg BID vs Placebo; Baseline is defined as the Day -2 assessment; Test type: Superiority or Other; p = 0.9810, ANCOVA; [statistical method as in outcome 6, analysis 2]; LSMean difference from placebo = -4.01, 92% CI 1-sided [lower limit -6.70], Standard Error of Mean 1.902

7. Primary Outcome: Change From Baseline in Blood Oxygen Level Dependent (BOLD) fMRI Activation Parameter Estimates (Z-scores) in Anterior Ventral Striatum Region of Interest (ROI) for the Contrast of Cue Gain > Cue No Gain in Monetary Incentive Delay (MID) Task on Day 15
Description: MRI parameter estimates refer to the 90th percentile Z-statistics across all voxels within the Region of Interest (ROI). This task provided a measure of reward anticipation and reward consummation. One of 3 shapes was presented on the screen (each uniquely associated with gain, loss and neutral) as a cue, and participants were instructed to respond to each cue, using their dominant hand, by pressing in response to a subsequent target that appeared for a variable length of time. Baseline was defined as Day 0 assessment. To be included in analysis participants must have complete Monetary Incentive Delay (MID) data at both Baseline and post-baseline, without excessive head motion. Participants with MID <40% at baseline were excluded from the analysis and summary statistics. Scores were not bounded by a minimum or maximum range, higher z-score implies a greater motivation of the participant by the prospect of monetary gain than no monetary gain.
Time Frame: Baseline, Day 15
Population: PPAS was used,defined as subset of FAS dataset.Criteria for PPAS:1)Received all doses of study treatment to which they were randomized;2)No major protocol deviation;3)Had a baseline measurement and at least 1 post baseline measurement for at least 1 PD endpoint.Overall Number of Participants Analyzed=participants evaluable in this outcome measure.
Measure: Mean (Standard Deviation); unit: Z scores
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Number analyzed (Participants) | 13 | 15 | 24 | 25
Z scores | 0.045 (1.092) | -0.229 (1.042) | 0.075 (1.139) | -0.048 (0.991)
Statistical Analysis 1: Comparison: PF-06412562 3 mg BID vs Placebo; Baseline is defined as the Day 0 assessment; Test type: Superiority or Other; p = 0.4821, ANCOVA; One (1)-side P-values were obtained from an ANCOVA model on change from baseline with baseline, treatment, site, gender and age as fixed effects; LSMean difference from placebo = 0.0129, 99% CI 1-sided [lower limit -0.6682], Standard Error of Mean 0.2860
Statistical Analysis 2: Comparison: PF-06412562 9 mg BID vs Placebo; Baseline is defined as the Day 0 assessment; Test type: Superiority or Other; p = 0.8576, ANCOVA; [statistical method as in outcome 7, analysis 1]; LSMean difference from placebo = -0.2974, 99% CI 1-sided [lower limit -0.9547], Standard Error of Mean 0.2760
Statistical Analysis 3: Comparison: PF-06412562 45 mg BID vs Placebo; Baseline is defined as the Day 0 assessment; Test type: Superiority or Other; p = 0.4182, ANCOVA; [statistical method as in outcome 6, analysis 2]; LSMean difference from placebo = 0.0498, 99% CI 1-sided [lower limit -0.5226], Standard Error of Mean 0.2403

8. Secondary Outcome: Plasma Concentrations of PF-06412562 for Each Dose.
Description: PF-06412562 plasma concentration for each dose at 6 and 12 hours on Days 1, 7 and 12, as well as 0 hours on Day 16.
Time Frame: 6, and 12 hours on Days 1, 7 and 12, as well as 0 hours on Day 16
Population: The PK concentration analysis set was defined as all participants randomized and treated who had at least 1 PK concentration. Here, "number analyzed" signifies the participants evaluable for each time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID
Number analyzed (Participants) | 22 | 16 | 33
ng/mL
  6h on Day 1: number analyzed (Participants) | 16 | 15 | 27
  6h on Day 1 | 19.99 (5.315) | 61.59 (26.366) | 100.9 (41.694)
  12h on Day 1 | 16.14 (5.8686) | 47.88 (18.211) | 79.67 (37.939)
  6h on Day 7: number analyzed (Participants) | 16 | 12 | 26
  6h on Day 7 | 44.89 (34.585) | 113.8 (44.331) | 581.1 (309.63)
  12h on Day 7: number analyzed (Participants) | 22 | 16 | 32
  12h on Day 7 | 29.65 (24.259) | 72.59 (31.865) | 365.3 (179.43)
  6h on Day 12: number analyzed (Participants) | 17 | 12 | 24
  6h on Day 12 | 33.47 (10.815) | 92.39 (44.805) | 533.2 (298.43)
  12h on Day 12: number analyzed (Participants) | 22 | 16 | 30
  12h on Day 12 | 25.34 (12.383) | 67.34 (36.958) | 357.0 (160.09)
  0h on Day 16: number analyzed (Participants) | 22 | 16 | 29
  0h on Day 16 | 17.14 (24.418) | 24.96 (17.571) | 164.9 (105.95)

9. Secondary Outcome: Plasma Concentrations of PF-06663872 at for Each Dose.
Description: PF-06412562 plasma concentration for each dose at times 6 and 12 hours on Days 1, 7 and 12, as well as 0 hours on Day 16.
Time Frame: 6 and 12 hours on Days 1, 7 and 12, as well as 0 hours on Day16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID
Number analyzed (Participants) | 22 | 16 | 33
ng/mL
  6h on Day 1: number analyzed (Participants) | 16 | 15 | 27
  6h on Day 1 | 1.707 (0.45216) | 5.649 (3.1174) | 8.894 (4.1986)
  12h on Day 1 | 1.948 (0.44567) | 5.355 (2.0234) | 8.108 (3.4277)
  6h on Day 7: number analyzed (Participants) | 16 | 12 | 26
  6h on Day 7 | 5.289 (4.6182) | 12.00 (3.3004) | 58.36 (22.666)
  12h on Day 7: number analyzed (Participants) | 22 | 16 | 32
  12h on Day 7 | 4.218 (4.9360) | 8.758 (3.3431) | 43.06 (16.824)
  6h on Day 12: number analyzed (Participants) | 17 | 12 | 24
  6h on Day 12 | 3.733 (1.1179) | 10.27 (4.9097) | 53.39 (24.715)
  12h on Day 12: number analyzed (Participants) | 22 | 16 | 30
  12h on Day 12 | 3.144 (0.95169) | 8.604 (4.2130) | 40.95 (14.892)
  0h on Day 16: number analyzed (Participants) | 22 | 16 | 29
  0h on Day 16 | 2.925 (4.8908) | 3.432 (2.1968) | 19.25 (9.0442)

ADVERSE EVENTS:
Time Frame: Baseline up to 7-10 days after last dose of study drug, up to 26 days
Arm/Group | PF-06412562 3 mg BID | PF-06412562 9 mg BID | PF-06412562 45 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/16 | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 7/22 | 10/16 | 17/33 | 12/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06412562 3 mg BID (N=22) | PF-06412562 9 mg BID (N=16) | PF-06412562 45 mg BID (N=33) | Placebo (N=29)
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06412562 3 mg BID (N=22) | PF-06412562 9 mg BID (N=16) | PF-06412562 45 mg BID (N=33) | Placebo (N=29)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 5 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 3 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 8 | 1
Sedation (Nervous system disorders) | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 4
Abnormal dreams (Psychiatric disorders) | 0 | 3 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.